CLINICAL TRIAL: NCT05952089
Title: An Open-label, Single-sequence Study to Evaluate the Effect of Coadministration of Danicamtiv on the Pharmacokinetics of Midazolam in Patients With Stable Heart Failure With Reduced Ejection Fraction
Brief Title: A Study to Assess the Effect of Danicamtiv on the Drug Levels of Midazolam in Participants With Stable Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV028-009
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: HFrEF; Danicamtiv; BMS-986434; MYK-491; Midazolam
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Danicamtiv + Midazolam (Experimental)
  Interventions: Drug: Danicamtiv; Drug: Midazolam

INTERVENTIONS:
Drug: Danicamtiv — Specified dose on specified days
  Other Names: BMS-986434; MYK-491
Drug: Midazolam — Specified dose on specified days

SUMMARY:
The purpose of this study is assess the effect of danicamtiv, as an inducer on the drug levels of midazolam in participants with heart failure with reduced ejection fraction (HFrEF).

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory participants with stable HFrEF due to any etiology.
* Body mass index (BMI) of 18.0 kilogram per square meter (kg/m2) to 35.0 kg/m2 inclusive.
* Documented left ventricular ejection fraction (LVEF) 15% to 45% (on 2 occasions), including at least once during Screening and confirmed by the Echo Core Laboratory (the absolute difference between the 2 LVEF values qualifying the participant should be < 12%).
* Participant receiving chronic medication for the treatment of heart failure reflecting current guidelines, including at least one of the following, unless not tolerated or contraindicated:β-blocker, angiotensin converting enzyme inhibitor, angiotensin receptor blocker, or angiotensin receptor neprilysin inhibitor. Such treatments should have been given at stable doses for at least ≥ 2 weeks prior to screening with no plan to modify treatments during the study.
* Sinus rhythm or stable atrial or ventricular pacing or persistent atrial fibrillation that is adequately rate-controlled to allow pharmacodynamic (PD) assessments by Transthoracic echocardiogram (TTE). NOTE: Participants with implanted cardioverter defibrillator (ICD), pacing, or cardiac resynchronization therapy are eligible provided device programming is unchanged starting 2 months prior to and throughout the dosing period.
* Adequate acoustic windows, determined by the Echo Core Laboratory, to enable accurate TTE assessments.

Exclusion Criteria:

* Presence of disqualifying cardiac rhythms that would preclude echocardiographic assessments, as determined by the Investigator, including: (a) rapid, inadequately rate controlled atrial fibrillation or (b) frequent premature ventricular contractions that might interfere with reliable echocardiographic measurements of left ventricular function.
* History of bronchospasm, or history of respiratory depression or arrest, airway obstruction, oxygen desaturation, or apnea.
* History of allergy to midazolam, other benzodiazepines, danicamtiv, related compounds, or excipients in the formulations.
* Severe renal insufficiency (defined as current estimated glomerular filtration rate [eGFR] < 30 mL/min/1.73 m2 by simplified Modification of Diet in Renal Disease equation [sMDRD].

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to Day 12
Area under the plasma concentration time curve from time zero extrapolated to infinite time (AUC[INF]) | Up to Day 12
Area under the plasma concentration time curve from time zero to the time of the last quantifiable concentration (AUC[0-T]) | Up to Day 12

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) | Up to Day 12
Terminal elimination half-life (T-HALF) | Up to Day 12
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to Day 12
Number of participants with vital sign abnormalities | Up to Day 12
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 12
Number of participants with physical examination abnormalities | Up to Day 12
Number of participants with clinical laboratory abnormalities | Up to Day 11

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (5):
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Research Integrity LLC, Owensboro, Kentucky
  - Sinai Hospital Of Baltimore, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome